CLINICAL TRIAL: NCT03853902
Title: MOSAIC-P: Mindfulness Online for Symptom Alleviation and Improvement in Cancer of the Prostate
Brief Title: Mindfulness Online for Symptom Alleviation and Improvement in Cancer of the Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Principal Investigator, David Victorson, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EH15-403
Record Dates: First submitted 2018-12-12; First posted 2019-02-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; mindfulness; MBSR; online course
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into a mindfulness course online or a mindfulness course in-person
Who Masked: Participant
Masking Description: Participants will not be told which is the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Program Online (Experimental): Online 4-week mindfulness program that is intended to reduce stress and improve the quality of life of patients with metastatic prostate cancer
  Interventions: Behavioral: Mindfulness Program
- Mindfulness Program Face-to-Face (Active Comparator): In-person 4-week mindfulness program that is intended to reduce stress and improve the quality of life of patients with metastatic prostate cancer
  Interventions: Behavioral: Mindfulness Program

INTERVENTIONS:
Behavioral: Mindfulness Program — Mindfulness Program

SUMMARY:
In this study, the researchers will examine the effects of a 4-week online mindfulness intervention, compared to a face-to-face mindfulness intervention, to reduce self-reported symptoms of fatigue, anxiety, depression, sleep disturbance, and pain interference in a sample of patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
Participants will be recruited from multiple locations, including NorthShore University Health System's Kellogg Cancer Center (KCC) and local community organizations (e.g., UsToo meetings, Cancer Wellness Center). Participating physician researchers will identify their eligible patients from the electronic medical record and will mail them a letter of invitation to learn more about the study and consider enrolling. Each participant will be e-mailed a link to the baseline questionnaire. After baseline completion, participants will be randomized, using an online random number generator, to the online course or face-to-face course. Course orientation for both groups will be held on the same night, but at different times. The separate orientations will be scheduled with a thirty minute break in between, in order to prevent intermixing of the groups and potential dissatisfaction among participants about their assigned group. In the orientation for the online class, participants will become familiar with the online video conferencing program Zoom, be introduced to other group participants, and receive a clear overview of what to expect for the 4-week mindfulness course. In the orientation for the face-to-face class, participants will be introduced to other group participants and receive a clear overview of what to expect for the 4-week mindfulness course. Participants will meet for approximately 2.5 hours each week for 4 weeks online or face-to-face. In addition, a face to face half day retreat will occur after the third class, in which participants from both face to face and online courses may attend. In the event that a participant unexpectedly misses a class, the instructor will follow-up with them and review the material covered in class. The class instructor may contact participants up to 3 times to review class expectations and teachings prior to or during the 4-week program. Participants will once again be asked to complete the online assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically advanced prostate cancer (e.g., castrate-sensitive, metastatic [clinical metastasis], castrate-resistant, non-metastatic [rising PSA on LHRH], castrate-resistant, metastatic)
* Receiving some form of cancer treatment (e.g., androgen deprivation therapy, chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-217
* At least 18 years of age
* Able to speak, read and understand English
* Able to perform basic activities of daily living (as determined by referring physician)
* Cognitively intact and free of serious psychiatric illness (as determined by referring physician)
* Access to internet connection within a room where patient will not be interrupted. This room needs to have an open space of about 6ft by 5 ft to allow for gentle movement and stretching.
* Access to a laptop or desktop computer with a camera. In the event that a patient does not have access to a computer, but is committed to the course, a laptop will be lent to him from the Department of Medical Social Sciences at Northwestern University.
* Willing to commit to the online MBSR course
* Willing to complete pre- and post-test assessments
* Physically able to participate in gentle Hatha yoga postures that are geared towards cancer patient populations, as determined by referring physician or medical team member

Exclusion Criteria:

* Regular user of MBSR or a similar mind-body therapy, which is defined as ≥ 4 times a week for the past 2 weeks
* Men with a short life expectancy as determined by the referring oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Change in pain interference using the PROMIS Pain Interference questionnaire | baseline, week 4
  Participants were administered the PROMIS Pain Interference questionnaire. The PROMIS Pain Interference measures the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. PROMIS Pain interference also incorporates items probing sleep and enjoyment in life, though it only contains one sleep item. The PROMIS Pain Interference is generic rather than disease-specific. It assesses pain interference over the past seven days. Each question has five response options ranging in value from one to five (1=not at all; 2=a little bit; 3=somewhat; 4=quite a bit; 5=very much). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. A higher score represents more of the concept being measured.
Change in sleep using the PROMIS Sleep Disturbance questionnaire | baseline, week 4
  Participants were administered the PROMIS Sleep Disturbance questionnaire. The PROMIS Sleep Disturbance assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. It does not focus on symptoms of specific sleep disorders, nor does it provide subjective estimates of sleep quantities. The PROMIS Sleep Disturbance is universal rather than disease-specific. It assesses sleep disturbance over the past seven days. Each question has five response options ranging in value from one to five (1=not at all; 2=a little bit; 3=somewhat; 4=quite a bit; 5=very much). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. A higher score represents more of the concept being measured.
Change in depression using the PROMIS Depression questionnaire | baseline, week 4
  Participants were administered the PROMIS Depression questionnaire. The PROMIS Depression assesses self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Somatic symptoms are not included, which eliminates consideration of these items' confounding effects when assessing patients with co-morbid physical conditions. The PROMIS Depression is universal rather than disease-specific. It assesses depression over the past seven days. Each question has five response options ranging in value from one to five (1=never; 2=rarely; 3=sometimes; 4=often; 5=always). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. A higher score represents more of the concept being measured.
Change in anxiety using the PROMIS Anxiety questionnaire | baseline, week 4
  Participants were administered the PROMIS Anxiety questionnaire. The PROMIS Anxiety measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Only one behavioral avoidance item is included; therefore, behavioral fear avoidance is not fully evaluated. The PROMIS Anxiety is universal rather than disease-specific. It assesses anxiety over the past seven days. Each question has five response options ranging in value from one to five (1=never; 2=rarely; 3=sometimes; 4=often; 5=always). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. A higher score represents more of the concept being measured.
Change in fatigue using the PROMIS Fatigue questionnaire | baseline, week 4
  Participants were administered the PROMIS Fatigue questionnaire. The PROMIS Fatigue evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities.The PROMIS Fatigue is universal rather than disease-specific. It assesses fatigue over the past seven days. Each question has five response options ranging in value from one to five (1=never; 2=rarely; 3=sometimes; 4=often; 5=always). To find the total raw score, sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. A higher score represents more of the concept being measured.

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Society AC. American Cancer Society Cancer Facts & Figures. Atlanta: American Cancer Society; 2014
- [Background] Resnick MJ, Penson DF. Quality of life with advanced metastatic prostate cancer. Urol Clin North Am. 2012 Nov;39(4):505-15. doi: 10.1016/j.ucl.2012.07.007. Epub 2012 Aug 27. PMID 23084527
- [Background] Sartor O, Flood E, Beusterien K, Park J, Webb I, MacLean D, Wong BJ, Mark Lin H. Health-related quality of life in advanced prostate cancer and its treatments: biochemical failure and metastatic disease populations. Clin Genitourin Cancer. 2015 Apr;13(2):101-12. doi: 10.1016/j.clgc.2014.08.001. Epub 2014 Aug 19. PMID 25262852
- [Background] Lengacher CA, Johnson-Mallard V, Barta M, Fitzgerald S, Moscoso MS, Post-White J, Jacobsen PB, Molinari Shelton M, Le N, Budhrani P, Goodman M, Kip KE. Feasibility of a mindfulness-based stress reduction program for early-stage breast cancer survivors. J Holist Nurs. 2011 Jun;29(2):107-17. doi: 10.1177/0898010110385938. Epub 2010 Nov 1. PMID 21041554
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868
- [Background] Bishop SR, Lau M, Shapiro S, et al. Mindfulness: A Proposed Ooperational Definition. Clinical Psychology: Science and Practice. 2004 2004;11(3):230-241
- [Background] Hulsheger UR, Alberts HJ, Feinholdt A, Lang JW. Benefits of mindfulness at work: the role of mindfulness in emotion regulation, emotional exhaustion, and job satisfaction. J Appl Psychol. 2013 Mar;98(2):310-25. doi: 10.1037/a0031313. Epub 2012 Dec 31. PMID 23276118
- [Background] Kabat-Zinn J. Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing; 1990
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003 Jul-Aug;65(4):571-81. doi: 10.1097/01.psy.0000074003.35911.41. PMID 12883107
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] Saxe GA, Major JM, Nguyen JY, Freeman KM, Downs TM, Salem CE. Potential attenuation of disease progression in recurrent prostate cancer with plant-based diet and stress reduction. Integr Cancer Ther. 2006 Sep;5(3):206-13. doi: 10.1177/1534735406292042. PMID 16880425
- [Background] Victorson D, Du H, Hankin V, et al. MINDFULNESS BASED STRESS REDUCTION DECREASES FEAR OF PROGRESSION OVER TIME FOR MEN WITH PROSTATE CANCER ON ACTIVE SURVEILLANCE: RESULTS FROM A RANDOMIZED CLINICAL TRIAL. The Journal of Urology. 2012 2012;187(4S):384
- [Background] Zernicke KA, Campbell TS, Speca M, McCabe-Ruff K, Flowers S, Dirkse DA, Carlson LE. The eCALM Trial-eTherapy for cancer appLying mindfulness: online mindfulness-based cancer recovery program for underserved individuals living with cancer in Alberta: protocol development for a randomized wait-list controlled clinical trial. BMC Complement Altern Med. 2013 Feb 16;13:34. doi: 10.1186/1472-6882-13-34. PMID 23414206
- [Background] Cavanagh K, Strauss C, Cicconi F, Griffiths N, Wyper A, Jones F. A randomised controlled trial of a brief online mindfulness-based intervention. Behav Res Ther. 2013 Sep;51(9):573-8. doi: 10.1016/j.brat.2013.06.003. Epub 2013 Jun 28. PMID 23872699
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Trapnell PD, Campbell JD. Private self-consciousness and the five-factor model of personality: distinguishing rumination from reflection. J Pers Soc Psychol. 1999 Feb;76(2):284-304. doi: 10.1037//0022-3514.76.2.284. PMID 10074710
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Rose M, Bjorner JB, Becker J, Fries JF, Ware JE. Evaluation of a preliminary physical function item bank supported the expected advantages of the Patient-Reported Outcomes Measurement Information System (PROMIS). J Clin Epidemiol. 2008 Jan;61(1):17-33. doi: 10.1016/j.jclinepi.2006.06.025. PMID 18083459
- [Background] Gershon R. Comparing short forms and CAT across PROMIS. 2009
- [Background] Roth AJ, Rosenfeld B, Kornblith AB, Gibson C, Scher HI, Curley-Smart T, Holland JC, Breitbart W. The memorial anxiety scale for prostate cancer: validation of a new scale to measure anxiety in men with with prostate cancer. Cancer. 2003 Jun 1;97(11):2910-8. doi: 10.1002/cncr.11386. PMID 12767107
- [Background] Lai J-S, Cella D, Choi S, Teresi JA, Hays RD, Stone AA. Developing a fatigue item bank for the Patient-Reported Outcomes Measurement Information System (PROMIS FIB version 1). Presented at the Meeting of the Survey Methods in Multicultural, Multinational, and Multiregional Contexts (3MC), Berlin, Germany. 2008
- [Background] Flynn KE, Shelby RA, Mitchell SA, Fawzy MR, Hardy NC, Husain AM, Keefe FJ, Krystal AD, Porter LS, Reeve BB, Weinfurt KP. Sleep-wake functioning along the cancer continuum: focus group results from the Patient-Reported Outcomes Measurement Information System (PROMIS((R))). Psychooncology. 2010 Oct;19(10):1086-93. doi: 10.1002/pon.1664. PMID 20013938
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116